CLINICAL TRIAL: NCT05431816
Title: Effect of Dietary Fiber Intervention on Patients With Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: M2021570
Record Dates: First submitted 2022-03-15; First posted 2022-06-24 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary fiber intervention (Experimental): Participants take a certain amount of dietary fiber per day.
  Interventions: Dietary Supplement: Dietary intervention
- Placebo (Placebo Comparator): Participants take a certain amount of placebo (Maltodextrin) per day.
  Interventions: Dietary Supplement: Dietary intervention

INTERVENTIONS:
Dietary Supplement: Dietary intervention — dietary fiber （Inulin 4g，Resistant Starch 4g，β-glucan 2g）

SUMMARY:
The purpose of the study is to understand the effect of dietary fiber on patients with polycystic ovary syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are 20 to 40 years old, planning to become pregnant or infertile women.
2. Individuals who are diagnosed as PCOS according to Rotterdam PCOS diagnostic criteria: 1）oligomenorrhea or amenorrhea or irregular uterine bleeding 2) hyperandrogenism or hyperandrogenism; 3) ultrasonography showing polycystic ovary, while excluding other diseases that may cause hyperandrogenism and ovulation abnormalities. Meets at least two of the three criterias.
3. Individuals who can insist on continuous monitoring in the outpatient clinic,
4. Individuals who are not participating in other research projects currently or 3 months before the intervention.

Exclusion Criteria:

1. Individuals who suffering from other diseases that may cause hyperandrogenism and ovulation abnormalities.
2. Individuals who are during pregnant, lactation or menopause.
3. Individuals who currently receiving weight-loss drugs or surgery or within the past 2 months.
4. Individuals who suffer from infectious diseases such as hepatitis B, active tuberculosis, AIDS, etc.
5. Individuals who need regular medication to treat chronic diseases such as diabetes, hypertension, gout, hyperuricemia, etc.
6. Use of medications that affect hormone levels, appetite, carbohydrate absorption, and metabolism within the past 2 months.
7. Individuals with severe liver diseases or kidney disease that are ineligible to participate in the study.
8. A medical history of severe cardiovascular and cerebrovascular diseases.
9. Individuals who currently suffer from severe gastrointestinal diseases or undergo gastrointestinal resection that may affect nutrient absorption.
10. Individuals who drink more than 15g of alcohol per day or have a smoking habit.
11. Individuals who need drug treatment for any mental illness such as epilepsy and depression.
12. Cancer patients.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota | before and after 2,4,8,12 weeks of intervention
  Study the gut microbiota change of stool samples between placebo group and intervention group
Changes in metabolomics | before and after 2,4,8,12 weeks of intervention
  Study the netabolomics change of stool samples between placebo group and intervention group
Changes in endocrine hormones | before and after 12 weeks of intervention
  Study the hormones change of blood samples between placebo group and intervention group
Changes in ovarian volume | before and after 12 weeks of intervention
  The size of each ovary will be determined using transvaginal ultrasonography for each participant in early follicular phase.
Changes in the number of follicles | before and after 12 weeks of intervention
  The number of follicles of each ovary will be determined using transvaginal ultrasonography for each participant in early follicular phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Patients' information is requested to be confidential.